CLINICAL TRIAL: NCT01773993
Title: SPECIAL INVESTIGATION OF PREGABALIN FOR FIBROMYALGIA
Brief Title: Special Investigation of Pregabalin for Fibromyalgia (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081282
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Pain Associated With Fibromyalgia
Keywords: Lyrica; pregabalin; Good post marketing practice; Post Marketing Surveillance; Regulatory Post Marketing Commitment Plan; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregabalin: Subjects who are treated with pregabalin
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — The usual adult dosage for oral use begins at 150 mg/day of pregabalin twice daily, and should be gradually increased to 300 mg/day over 1 week or more and then maintained at 300-450 mg/day as needed. Dosage should be adjusted, depending on age or symptoms. However, the daily maximum dose should not be beyond 450 mg, and should be orally administered twice daily.
  Other Names: Lyrica® Capsules 25 mg, Lyrica® Capsules 75 mg, Lyrica® Capsules 150 mg

SUMMARY:
To collect the efficacy and safety information of Pregabalin on Fibromyalgia patients related to their appropriate use in daily practice.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first pregabalin should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Fibromyalgia
* Pregabalin naive patient

Exclusion Criteria:

* Clinical diagnosis of neuropathic pain

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic and hospital for Fibromyalgia
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081282&StudyName=Special%20Investigation%20of%20Pregabalin%20for%20Fibromyalgia%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- LYRICA Capsules (Pregabalin): Participants who received LYRICA Capsules as indicated in the approved local product document were observed for a period of 52 weeks at maximum. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | LYRICA Capsules (Pregabalin)
Started | 534
Completed | 499 (Number of participants whose survey form were collected and included in analyses is shown.)
Not Completed | 35
Not completed — No Visit After Treatment | 35

BASELINE CHARACTERISTICS:
Population: Among 534 participants whose survey form was collected, a total of 35 participants were excluded from the baseline analysis population due to no visit after treatment.
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Age, Customized [Number; unit: Participants]
  <15 years | 1
  ≥15 and <65 years | 392
  ≥65 years | 106
Sex/Gender, Customized [Number; unit: Participants]
  Male | 91
  Female | 408
Race/Ethnicity, Customized [Number; unit: Participants]
  Race and Ethnicity Not Collected | 499

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to 52 weeks at maximum
Population: The analysis population for this outcome measure was the baseline analysis population, which comprised of participants who satisfied the criteria of safety analysis population and had received LYRICA Capsules at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Percentage of Participants | 25.45

2. Secondary Outcome: Percentage of Participants With Serious Adverse Drug Reaction
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Percentage of Participants | 0.20

3. Secondary Outcome: Percentage of Participants With Adverse Drug Reaction Unexpected From Japanese Package Insert
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to LYRICA Capsules was assessed by the physician.
Time Frame: From Week 1 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Percentage of Participants | 3.41

4. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Peripheral Edema or Other Edema-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to peripheral edema or other edema-related events was evaluated.
Time Frame: From Week 1 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Participants | 6

5. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Dizziness, Somnolence, Loss of Consciousness, Syncope, and Potential for Accidental Injury
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to dizziness, somnolence, loss of consciousness, syncope, and potential for accidental injury was evaluated.
Time Frame: From Week 1 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Participants | 65

6. Secondary Outcome: Number of Participants With Adverse Drug Reactions Related to Vision-related Events
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to LYRICA Capsules in a participant who received LYRICA Capsules. Relatedness to LYRICA Capsules was assessed by the physician. Occurrence of ADRs related to vision-related events was evaluated.
Time Frame: From Week 1 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 499
Participants | 5

7. Secondary Outcome: Change From Baseline in Pain Score at Week 52
Description: The pain from fibromyalgia experienced during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (no pain) to 10 (the most severe pain possible). Mean change from baseline in the pain score at Week 52 was presented along with standard deviation.
Time Frame: Baseline and at Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of pain score was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 182
Units on a scale | -2.4 (2.67)

8. Secondary Outcome: Change From Baseline in Quality of Sleep Score at Week 52
Description: The quality of sleep experienced during the past 24 hours was rated by participants at the time of getting up in the morning on an 11-grade scale, ranging from 0 (the best sleep possible) to 10 (the worst sleep possible). Mean change from baseline in quality of sleep score at Week 52 was presented along with standard deviation.
Time Frame: Baseline and at Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of quality of sleep score was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 163
Units on a scale | -1.4 (2.71)

9. Secondary Outcome: Patient's Impression (PGIC) at Week 52
Description: The patient's impression (patient global impression of change [PGIC]) at Week 52, as compared to the baseline condition (including the first day of treatment), was rated by participants on a 7-grade scale.
Time Frame: At Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of PGIC was available among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 416
Participants
  Markedly improved | 34
  Improved | 79
  Slightly improved | 119
  Unchanged | 65
  Slightly worsened | 6
  Worsened | 3
  Markedly worsened | 1
  Not assessed | 109

10. Secondary Outcome: Physician's Impression (CGIC) at Week 52
Description: The physician's impression (clinical global impression of change [CGIC]) at Week 52, as compared to the baseline condition (including the first day of treatment), was rated by the physician on a 7-grade scale.
Time Frame: At Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of CGIC was available among the baseline analysis population.
Measure: Number; unit: Participants
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 409
Participants
  Markedly improved | 45
  Improved | 105
  Slightly improved | 121
  Unchanged | 59
  Slightly worsened | 4
  Worsened | 2
  Markedly worsened | 1
  Not assessed | 72

11. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Score at Week 52
Description: The problems associated with depression-related symptoms experienced during the last 2 weeks were rated by participants ranging from 0 (not at all) to 3 (nearly every day) in total 0 to 27(the higher the more severe) consisting the following 9 items: 1) little interest or pleasure in doing things; 2) depressed, or hopeless; 3) trouble falling or staying asleep, or sleeping too much; 4) feeling tired or having little energy; 5) poor appetite or overeating; 6) feeling bad about yourself - or that you are a failure or have let yourself or your family down; 7) trouble concentrating on things, such as reading the newspaper or watching television; 8) moving or speaking so slowly that other people could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual; and 9) thoughts that you would be better off dead, or of hurting yourself. Mean change from baseline in the evaluation score was presented along with standard deviation.
Time Frame: Baseline and at Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of PHQ-9 was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 161
Units on a scale | -3.4 (6.91)

12. Secondary Outcome: Change From Baseline in Health Status of EuroQol 5 Dimension (EQ-5D) at 52 Weeks
Description: Health status (EQ-5D) was evaluated based on the following 5 dimensions: mobility, self-care, usual activity (e.g., work, study, housework, family, or leisure activities), pain/discomfort, and anxiety/depression. Each dimension was rated in the three levels of response alternatives "no problems," "some problems," or "extreme problems." For the analysis of EQ-5D, the response outcome for the five dimensions was converted to a utility value using tariff value set based on the Japanese version of EQ-5D. The utility value was not assigned if there was no response in any one of the five dimensions. 1 for full health and 0 for being dead: a positive (negative) number implies that the health state is better (worse) than dead. Mean change from baseline in the evaluation score was presented along with standard deviation.
Time Frame: Baseline and at Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of EQ-5D was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 162
Units on a scale | 0.1 (0.19)

13. Secondary Outcome: Change From Baseline in Fibromyalgia Activity Score (FAS-31) at 52 Weeks
Description: FAS-31 (ranged from 0 to 31) is calculated as the combined score of the widespread pain index (WPI, ranged from 0 to 19) and the symptom severity (SS) scale (ranged from 0 to 12). The WPI is a measure of the number of painful body regions. The SS is the scale of the severity in the three symptoms (fatigue, waking unrefreshed, and cognitive symptoms; ranged from 0 to 3 each) and general physical symptoms (ranged from 0 to 3). WPI ranged from 0 to 19 the higher score indicates more severe of activity, SS ranged from 0-12 also higher score shows more severe symptoms observed. Mean change from baseline in the evaluation score was presented along with standard deviation.
Time Frame: At Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of FAS-31 was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 175
Units on a scale | -5.2 (6.15)

14. Secondary Outcome: Change From Baseline in the Japanese Version of the Revised Fibromyalgia Impact Questionnaire (JFIQR) at 52 Weeks
Description: JFIQR is a Japanese version of the Revised Fibromyalgia Impact Questionnaire (FIQR), which was established for overall evaluation of the influence of fibromyalgia on patient's health. It consists of three linked sets of domains: "function (9 questions)," "overall impact (2 questions)," and "symptoms (10 questions)." Participants responded to the questions based on an 11-grade scale, ranging from 0 to 10, with 10 being the worst. For the analysis of JFIQR, the score for each domain was modified as follows: The summed score for "function" (ranged from 0 to 90) was divided by 3 and the summed score for "symptoms" (ranged from 0 to 100) was divided by 2. The summed score for "overall impact" (ranged from 0 to 20) was not modified. The total score, the sum of the three modified domain scores (ranged from 0 to 100, the lower score represents a better outcome), was used for the analysis. Mean change from baseline in the evaluation score was presented along with standard deviation.
Time Frame: At Week 52
Population: The analysis population for this outcome measure comprised of participants for whom the evaluation outcome of JFIQR was available among the baseline analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LYRICA Capsules (Pregabalin)
Number analyzed (Participants) | 137
Units on a scale | -15.2 (23.18)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | LYRICA Capsules (Pregabalin)
All-Cause Mortality (participants affected / at risk) | 0/499
Serious Adverse Events (participants affected / at risk) | 4/499
Other Adverse Events (participants affected / at risk) | 152/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=499)
Pneumonia bacterial (Infections and infestations) | 1
Loss of consciousness (Nervous system disorders) | 1
Angina unstable (Cardiac disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYRICA Capsules (Pregabalin) (N=499)
Anaemia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 2
Meniere's disease (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperprolactinaemia (Endocrine disorders) | 1
Foreign body sensation in eyes (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Lip blister (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 1
Discomfort (General disorders) | 1
Feeling abnormal (General disorders) | 3
Feeling cold (General disorders) | 1
Malaise (General disorders) | 3
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 8
Bronchitis (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia chlamydial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Lipids abnormal (Investigations) | 1
Weight increased (Investigations) | 18
Decreased appetite (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 38
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Restless legs syndrome (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 38
Affect lability (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Anxiety disorder (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 8
Mania (Psychiatric disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT01773993/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT01773993/SAP_001.pdf